CLINICAL TRIAL: NCT02360072
Title: To Delineate the Characteristics of Airway Inflammation and Bronchial Hyperresponsiveness in Rhinitic Children With or Without Asthma and Sought to Explore a Possible Predictor in the Progression of Allergic Rhinitis to Asthma
Brief Title: Airway Inflammation and Bronchial Hyperresponsiveness in Rhinitic Children With or Without Asthma
Status: Completed | Type: Observational
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, LI-HONG SUN, Professor, Guangzhou Institute of Respiratory Disease
Other Study IDs: GuangzhouIRD-LSUN1
Record Dates: First submitted 2015-02-05; First posted 2015-02-10 (Estimated); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Rhinitis; Asthma; Inflammation; Hypersensitivity
Keywords: child; allergic rhinitis; asthma; nitric oxide; bronchial hyper-responsiveness
MeSH Terms: conditions — Rhinitis; Asthma; Inflammation; Hypersensitivity; Rhinitis, Allergic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum ,nasal lavage fluid ,induced sputum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- AR group: Allergic rhinitis without any typical asthma symptoms
- Asthma: Accompanied by typical asthma symptoms and Δ FEV1≥12% in response to a short-acting bronchodilator or bronchial hyperreactivity(BHR) in the methacholine provocation test (PC20≤2.504mg)
- AR+Asthma: Diagnosed allergic rhinitis concomitant asthma symptoms
- Control group: non-atopic subjects with neither a history of rhinitis nor asthma

SUMMARY:
This is a prospective observational study , to clarity the characteristics of airway inflammation, airway reactivity and airway resistance in rhinitic children with or without asthma and to explore the possible predictors in the progression of allergic rhinitis to asthma.

DETAILED DESCRIPTION:
Children 6-15 years old with allergic rhinitis and/or asthma diagnosed by specialist physician are enrolled in the department of respiratory and otorhinolaryngology and pediatrics in Guangzhou Institute of Respiratory Disease. According to presence of typical symptoms and signs, patients are divided into allergic rhinitis without asthma (AR group) , allergic rhinitis concomitant asthma (AS+AR group), asthma without rhinitis (AS group). In addition, healthy students in a school are enrolled as normal control group. History of all subjects are collected, the following measurements are performed: skin prick test (SPT), peripheral blood cells five-classification test, serum total immunoglobulin E (IgE) and specific IgE of common inhalant allergens testing, nasal lavage and induced sputum cells classification ，pulmonary function test, bronchial provocation test using methacholine，airway resistance measured by impulse oscillation technique, the levels of eosinophil（ECP），eosinophil peroxidase（EPO）.Meanwhile myeloperoxidase （MPO）and eosinophil-derived neurotoxin (EDN) are measured in induced sputum ,in nasal lavage and in serum.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of allergic rhinitis and/or asthma
* Sensitized to more than 1 common aeroallergens

Exclusion Criteria:

* Respiratory infection 2 weeks prior to initial visit
* Children with nasal polyposis
* History of immunotherapy
* Unable to complete the test or had limited understanding
* Use of systemic corticosteroids 4 weeks prior to initial visit
* Nasal and inhaled corticosteroids 2 weeks prior to initial visit
* Leukotriene receptor antagonists 2 weeks prior to initial visit

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children 6-15 years old with allergic rhinitis and/or asthma diagnosed by specialist physician were enrolled in the department of paediatrics,respiratory and otorhinolaryngology in Guangzhou Institue of Respiratory Diseas .In addition, healthy students in a school were enrolled as normal control group.
Sampling Method: Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
To explore if an elevated level of fractional exhaled nitric oxide(FeNO) is a possible predictor of bronchial hyperresponsiveness in AR. | 1 year

SECONDARY OUTCOMES:
To explore if an elevated eosinophils in induced sputum is a possible predictor of bronchial hyperresponsiveness in AR. | 1 year
To explore if an elevated eosinophils in nasal nasal lavage fluid is a possible predictor of bronchial hyperresponsiveness in AR. | 1 year
To compare lower airway resistance (Z5,R5,X5,R5-20,R20 and Fres) using impulse oscillation among the groups [Allergic rhinitis(AR) group, Asthma group, AR+Asthma and control group]. | 1 year
To compare cumulative dosage of methacholine causing a 20% fall in forced expiratory volume in 1 second (PC20FEV1-MCH) among the groups. | 1 year
To compare forced vital capacity (FVC) , forced expiratory volume in 1 second (FEV1)， forced expired flow at 25% of FVC(FEF25) and forced expired flow at 75% of FVC (FEF75) among groups. | 1 year
To compare levels of eosinophil（ECP），eosinophil peroxidase（EPO）, myeloperoxidase （MPO）and eosinophil-derived neurotoxin (EDN) in induced sputum and nasal lavage fluid among the groups. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Nanshan Zhong, master, Study Director — Guangzhou Institute of Respiratory Disease
Locations (1):
- Guangzhou institute of respiratory disease, Guangzhou, Guangdong, China